CLINICAL TRIAL: NCT00044512
Title: A Phase II Multicenter Uncontrolled Trial of Sorafenib (BAY43-9006) in Patients With Advanced Hepatocellular Carcinoma
Brief Title: A Study to Estimate Safety and Efficacy of Sorafenib (BAY43-9006) in the Treatment of Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10874; NCT00048919 (obsolete NCT alias); NCT00058383 (obsolete NCT alias)
Record Dates: First submitted 2002-08-30; First posted 2002-09-04 (Estimated); Results first posted 2009-08-06 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-03

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Cancer; Liver Cancer; Hepatocellular carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasms; Liver Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sorafenib 400 mg b.i.d. (Experimental): Sorafenib (Nexavar, BAY43-9006) 400 mg administered bis in die (bid, twice a day)
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Sorafenib (Nexavar, BAY43-9006) 400 mg administered bis in die (bid, twice a day)

SUMMARY:
Evaluate anti-cancer activity (e.g. proportion of patients with confirmed complete response or partial response) in patients with advanced, inoperable biopsy-proven hepatocellular carcinoma.

DETAILED DESCRIPTION:
In addition to the key secondary outcome parameters the following exploratory parameters were evaluated in subpopulations:

* Pharmacokinetics (PK) profile of Sorafenib
* Plasma and tissue tumor biomarkers

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed primary hepatocellular carcinoma (HCC)
* Inoperable disease (T2-T4, any N, M0 or M1) or refused surgery
* Measurable disease
* At least 1 bidimensionally measurable lesion of at least 2 cm by computed tomography (CT) scan or magnetic resonance imaging (MRI)
* Presence of at least 1 of the following:
* Alpha-fetoprotein greater than the upper limit of normal (ULN)
* Hepatitis C antibody positive
* Hepatitis B surface antigen positive
* Child's Pugh class A or B
* Candidate for systemic therapy

Exclusion Criteria:

* Fibrolamellar disease mixed histology
* Metastatic brain or meningeal tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2002-08; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (21):
- United States (2):
  - Los Angeles, California
  - New York, New York
- Belgium (3):
  - Bruxelles - Brussel
  - Ghent
  - Leuven
- France (5):
  - Lille
  - Marseille
  - Paris
  - Rennes
  - Saint-Herblain
- Israel (6):
  - Haifa, Israel
  - Jerusalem, Israel
  - Petah Tikva, Israel
  - Rehovot, Israel
  - Tel Aviv, Israel
  - Tel Litwinsky
- Italy (5):
  - Rozzano, Milano
  - Forlì
  - Milan
  - Pisa
  - Verona

REFERENCES:
- [Result] Abou-Alfa GK, Schwartz L, Ricci S, Amadori D, Santoro A, Figer A, De Greve J, Douillard JY, Lathia C, Schwartz B, Taylor I, Moscovici M, Saltz LB. Phase II study of sorafenib in patients with advanced hepatocellular carcinoma. J Clin Oncol. 2006 Sep 10;24(26):4293-300. doi: 10.1200/JCO.2005.01.3441. Epub 2006 Aug 14. PMID 16908937
- [Result] Abou-Alfa GK, Amadori D, Santoro A, Figer A, De Greve J, Lathia C, Voliotis D, Anderson S, Moscovici M, Ricci S. Safety and Efficacy of Sorafenib in Patients with Hepatocellular Carcinoma (HCC) and Child-Pugh A versus B Cirrhosis. Gastrointest Cancer Res. 2011 Mar;4(2):40-4. PMID 21673874

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only subjects with measurable, histologically or cytologically documented hepatocellur carcinoma (HCC) which was inoperable or who had refused surgery could participate in this study.
Pre-assignment Details: Of 147 enrolled patients, 137 received treatment. 10 patients failed screening; reasons were: target lesions identified at baseline (3), liver function tests too high for inclusion (2), prior systemic anticancer treatment (2), creatinine too high for inclusion (1), platelets too low for inclusion (1), diagnosis of HCC not confirmed (1)
Period: Treatment
Arm/Group | Sorafenib 400 mg b.i.d.
Started | 137
Completed | 137
Not Completed | 0
Period: Follow Up
Arm/Group | Sorafenib 400 mg b.i.d.
Started | 137
Completed | 135
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Sorafenib 400 mg b.i.d.
Number analyzed (Participants) | 137
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 84
  >=65 years | 53
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 97
Child Pugh Status [Number; unit: participants] — A Child-Pugh (CP) score (determined by encephalopathy grade, ascites, serum bilirubin and albumin, prothrombin time) is used to assess the prognosis of chronic liver disease, mainly cirrhosis. One of the inclusion criterion for this study was a CP class A (good operative risk) or B (moderate risk) score; class C (poor operative risk) was excluded.
  participants
    Status A | 98
    Status B | 38
    Missing | 1
Eastern Cooperative Group performance status (ECOG PS) at study entry [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is a scale that measures how cancer affects a patient. 0 = fully active, 1 = restricted strenuous activity, 2 = ambulatory, 3 = limited selfcare, 4 = completely disabled, 5 = dead. Subjects entering this study must have had an ECOG score of 0 or 1.
  participants
    Grade 0 | 68
    Grade 1 | 69
    Grade 2 | 0
    Grade 3 | 0
    Grade 4 | 0
Stage of Disease at study entry (TNM Classification) [Number; unit: participants] — TNM (Tumor, Nodes, Metastasis) is a solid tumor classification system. T1-T4 = size and degree of spreading. N0-N3 = degree of spreading into lymph nodes. M0-M1 = whether the cancer has metastazied beyond the lymph nodes or not. Bigger numbers are worse. One of the inclusion criteria for this study was inoperable tumor T2-T4, any N, M0 or M1.
  participants
    Stage 1 | 0
    Stage 2 | 4
    Stage 3 | 42
    Stage 4 | 91

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants for Each Type of Response
Description: Objective response rate of sorafenib assessed as the proportion of subjects with confirmed complete or partial response as per modified World Health Organization (WHO) criteria.
Time Frame: Until 30 days after termination of active therapy
Population: Intention to Treat (ITT) analyses were performed on subgroups of patients categorized by baseline characteristics of ECOG Performance Status, Child Pugh status, TNM stage at study entry, prior surgical procedure, hepatitis A and B status, and age.
Measure: Number; unit: percentage of participants
Arm/Group | Sorafenib 400 mg b.i.d.
Number analyzed (Participants) | 137
percentage of participants
  Complete response (CR) | 0
  Partial response (PR) | 2.2
  Minor response (MR) | 5.8
  Stable disease (SD) | 54.7
  Progressive disease (PD) | 13.9
  Not available for independent review (NA) | 22.6
  Not evaluable (NE) | 0.7

2. Secondary Outcome: Duration of Response
Description: Duration of response was calculated from the first drug treatment date until documented progressive disease (PD). PD was 1) 25% or more increase in the sum of all target lesion areas taking as reference the smallest sum recorded at or following baseline, 2) unequivocal progression of an existing non-target lesion, or 3) appearance of a new lesion.
Time Frame: up to 3 years later
Population: Intention to Treat (ITT) analyses were performed on all treated subjects and for subgroups baseline Child Pugh status (A vs B), ECOG PS (0 vs 1), TNM stage at study entry (II/III vs IV), hepatitis B and C status (positive vs negative). The 3 subjects are censored at time of evaluation. The Median is not estimable so the reported number is biased.
Measure: Median (Full Range); unit: days
Arm/Group | Sorafenib 400 mg b.i.d.
Number analyzed (Participants) | 3
days | 374 [369 to 443]

3. Secondary Outcome: Time to Response
Description: Time from the first day of receiving study drug to the date the CR or PR was documented (with confirmation).
Time Frame: up to 3 years later
Population: Intention to Treat (ITT) analyses were performed on all treated subjects and for subgroups such as baseline Child Pugh status (A vs B), ECOG PS (0 vs 1), TNM stage at study entry (II/III vs IV), hepatitis B and hepatitis C status (positive vs negative).
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib 400 mg b.i.d.
Number analyzed (Participants) | 3
days | 144 [109 to 245]

4. Secondary Outcome: Time to Progression
Description: Time from the first date of receiving study drug until the first documented PD.
Time Frame: up to 3 years later
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib 400 mg b.i.d.
Number analyzed (Participants) | 106
days | 167 [140 to 284]

5. Secondary Outcome: Duration of Stable Disease
Description: Time from the first day of receiving study drug until there was a documented PD or response.
Time Frame: up to 3 years later
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib 400 mg b.i.d.
Number analyzed (Participants) | 103
days | 166 [135 to 275]

6. Secondary Outcome: Time to Minor Response
Description: Time from the first day of receiving study drug to the date the MR was first documented (with confirmation). Minor response = >25% regression.
Time Frame: up to 3 years later
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib 400 mg b.i.d.
Number analyzed (Participants) | 8
days | 84 [54 to 168]

7. Secondary Outcome: Duration of Minor Response
Description: Time from the date that MR was first documented to the date that PD was first documented.
Time Frame: Time from MR to PD
Population: as for outcome 3
Measure: Mean (Full Range); unit: days
Arm/Group | Sorafenib 400 mg b.i.d.
Number analyzed (Participants) | 8
days | 122 [49 to 222]

8. Secondary Outcome: Overall Survival
Description: Time from the first date of receiving study medication to death.
Time Frame: Start of treatment to death
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib 400 mg b.i.d.
Number analyzed (Participants) | 137
days | 280 [212 to 340]

ADVERSE EVENTS:
Description: Acronyms in Adverse Event section: Gastrointestinal (GI), Central Nervous System (CNS), Not Otherwise Specified (NOS), Absolute Neutrophil Count (ANC), Alanine Transaminase (ALT), Aspartate Transaminase (AST), Gamma Glutamyl Transpeptidase (GGT), Acute Respiratory Distress Syndrome (ARDS), Without grade 3 or 4 (W/O GR 3 or 4), Neutropenia (Neu)
Groups:
- Sorafenib 400 mg b.i.d.: Sorafenib (Nexavar, BAY43-9006) 400 mg administered b.i.d."Other AE" section includes SAEs
Arm/Group | Sorafenib 400 mg b.i.d.
Serious Adverse Events (participants affected / at risk) | 77/137
Other Adverse Events (participants affected / at risk) | 126/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib 400 mg b.i.d. (N=137)
Neutrophils (Blood and lymphatic system disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 6
Lymphopenia (Blood and lymphatic system disorders) | 1
Platelets (Blood and lymphatic system disorders) | 1
Supraventricular Arrythmia, Sinus Bradicardia (Cardiac disorders) | 1
Supraventricular Arrythmia, Supraventricular Tachycardia (Cardiac disorders) | 2
Hypertension (Cardiac disorders) | 1
Cardiac Ischemia / Infarction (Cardiac disorders) | 1
Hypotension (Cardiac disorders) | 3
Cardiac General - Other (Specify) (Cardiac disorders) | 1
Fever (General disorders) | 4
Fatigue (General disorders) | 9
Constitutional Symptoms - Other (Specify) (General disorders) | 4
Anorexia (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 4
Dehydration (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
GI - Other (Specify) (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Proctitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Hypercreatininemia (Renal and urinary disorders) | 1
Renal Failure (Renal and urinary disorders) | 3
Genito-Urinary - Other (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 2
CNS Hemorrhage (Vascular disorders) | 3
Melena / GI Bleeding (Vascular disorders) | 2
Epistaxis (Vascular disorders) | 1
Hemorrhage with Surgery (Vascular disorders) | 1
Hemorrhage - Other (Specify) (Vascular disorders) | 1
Rectal Bleeding (Vascular disorders) | 2
Hematuria (Vascular disorders) | 1
Hematemesis (Vascular disorders) | 6
Hemorrhage / Bleeding W/O GR 3 or GR 4 Thrombo (Vascular disorders) | 1
Hypoalbuminemia (Gastrointestinal disorders) | 1
Alkaline Phospharase (Hepatobiliary disorders) | 2
AST (Hepatobiliary disorders) | 1
Hyperbilirubinemia (Hepatobiliary disorders) | 8
Liver Dysfunction (Hepatobiliary disorders) | 15
GGT increase (Hepatobiliary disorders) | 1
Hepatobiliary - Other (Specify) (Hepatobiliary disorders) | 20
Infection W/GR 3 or GR 4 Neu (Infections and infestations) | 1
Infection without Neutropenia (Infections and infestations) | 9
Infection - Other (Specify) (Infections and infestations) | 1
Lymphatics - Other (Specify) (Blood and lymphatic system disorders) | 1
Musculoskeletal - Other (Specify) (Musculoskeletal and connective tissue disorders) | 3
Amylase (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypoglycemia (Metabolism and nutrition disorders) | 1
Lipase (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
CNS Ischemia (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 4
Dizziness (Nervous system disorders) | 1
Memory Impairment (Nervous system disorders) | 1
Neurology - Other (Specify) (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Syncope (Fainting) (Nervous system disorders) | 1
Glaucoma (Eye disorders) | 1
Chest Pain (General disorders) | 3
Pain, Abdomen NOS (General disorders) | 3
Pain - Other (Specify) (General disorders) | 3
ARDS (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary - Other (Specify) (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Shortness of Breath) (Respiratory, thoracic and mediastinal disorders) | 4
Head-Foot Skin Reaction (Skin and subcutaneous tissue disorders) | 2
Wound Complication, non-infectious (Skin and subcutaneous tissue disorders) | 1
Dermatology - Other (Specify) (Skin and subcutaneous tissue disorders) | 1
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib 400 mg b.i.d. (N=137)
Fatigue (General disorders) | 76
Anorexia (Gastrointestinal disorders) | 34
Diarrhea (Gastrointestinal disorders) | 76
Nausea (Gastrointestinal disorders) | 33
AST (Hepatobiliary disorders) | 28
Bilirubin (Hyperbilirubinemia) (Hepatobiliary disorders) | 40
Pain, Abdomen NOS (General disorders) | 49
Pain, Other (General disorders) | 32
Hand-Foot Skin Reaction (Skin and subcutaneous tissue disorders) | 42
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 29
Hemoglobin (Blood and lymphatic system disorders) | 14
Lymphopenia (Blood and lymphatic system disorders) | 8
Platelets (Blood and lymphatic system disorders) | 12
Edema (Cardiac disorders) | 21
Hypertension (Cardiac disorders) | 10
Fever (General disorders) | 18
Weight Loss (General disorders) | 13
Ascites (Gastrointestinal disorders) | 14
Constipation (Gastrointestinal disorders) | 26
GI-Other (Gastrointestinal disorders) | 21
Mucositis (Gastrointestinal disorders) | 19
Vomiting (Gastrointestinal disorders) | 26
Hypoalbuminemia (Hepatobiliary disorders) | 7
Alkaline Phosphatase (Hepatobiliary disorders) | 19
ALT (Hepatobiliary disorders) | 20
GGT (Hepatobiliary disorders) | 13
Hepatobiliary-Other (Hepatobiliary disorders) | 8
Infection Without Neutropenia (Infections and infestations) | 20
Amylase (Metabolism and nutrition disorders) | 9
Hyperglycemia (Metabolism and nutrition disorders) | 7
Lipase (Metabolism and nutrition disorders) | 10
Metabolic/Lab-Other (Metabolism and nutrition disorders) | 14
Dizziness (Nervous system disorders) | 11
Pain, Head/Headache (General disorders) | 11
Pain, Muscle (General disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 15
Pulmonary-Other (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnea (Shortness of Breath) (Respiratory, thoracic and mediastinal disorders) | 16
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 7
Alopecia (Skin and subcutaneous tissue disorders) | 16
Dermatology-Other (Skin and subcutaneous tissue disorders) | 12
Pruritus (Skin and subcutaneous tissue disorders) | 15

LIMITATIONS AND CAVEATS:
Subjects had advanced disease and were heavily pretreated. National Cancer Institute-Common Toxicity Criteria (NCI-CTC) was translated to Medical Dictionary for Regulatory Activities (MedDRA) for System Organ Class (SOC) only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreement between Sponsor and PI should be reached before publication